CLINICAL TRIAL: NCT02469220
Title: Diet Treatment of Patients With Ulcerative Colitis in Remission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regionshospital Nordjylland (Other Government)
Responsible Party: Principal Investigator, Anne Lund Krarup, MD, PhD, Regionshospital Nordjylland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RHN_ALK_01
Record Dates: First submitted 2015-06-08; First posted 2015-06-11 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Ulcerative Colitis
Keywords: Diet; low FODMAP; UC; IBS
MeSH Terms: conditions — Colitis, Ulcerative | interventions — FODMAP Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low FODMAP diet (Experimental): Diet with a low content of fermentable oligo-, di-, monosaccharides and polyols (low FODMAP diet). The patients will receive dietary instructions from registered clinical dieticians. A food supplement low in FODMAPS are administered in a blinded fashion.
  Interventions: Dietary Supplement: Low FODMAP
- Standardized FODMAP (Active Comparator): Diet with a low content of fermentable oligo-, di-, monosaccharides and polyols (low FODMAP diet). The patients will receive dietary instructions from registered clinical dieticians. A food supplement with FODMAPS are administered in a blinded fashion.
  Interventions: Dietary Supplement: Standardized FODMAP
- Control (No Intervention): Watchful waiting. No diets or food supplements are administered

INTERVENTIONS:
Dietary Supplement: Low FODMAP — Blinded food supplements containing only items with a low content of FODMAPs
  Arms: Low FODMAP diet
Dietary Supplement: Standardized FODMAP — Blinded food supplements containing FODMAPs
  Arms: Standardized FODMAP

SUMMARY:
The study examines the effect of a low FODMAP diet in patients with UC in remission but still having GI symptoms (IBS in IBD). 15 patients will be on watchful waiting. 15 patients will be on low FODMAP diet. 15 patients with recieve FODMAPs in their diet.

DETAILED DESCRIPTION:
Patients are randomized to either standard care, low FODMAP diet or a normal FODMAP diet. Run-in on a low FODMAP diet, thereafter parallel design where one arm is assign a blinded food supplement with low FODMAP content and the other arm is assigned a blinded food supplement containing FODMAP. A control group is "watchful waiting".

Symptom reports, blood, and fecal samples are collected.

ELIGIBILITY:
Inclusion Criteria:

* Colitis ulcerosa in remission (calciprotectin<200 and normal sigmoidoscopy)
* ROM IV criteria fullfilled
* Stable medical therapy

Exclusion Criteria:

* Intake of a low FODMAP diet within the past 6 weeks prior to baseline
* Atypical colitis ulcerosa primarily right sided disease and calciprotectin >50 unless normal sigmoidoscopy
* If diarrhea: Clostridium difficile infection
* Lactose intolerance
* Systemisk or local treatment for CU other than 5-aminosalicylicacid or biological therapy
* Antibiotics within 6 weeks
* Pregnancy
* Activity in UC
* Coeliac disease
* Abnormal transglutaminase
* Eating disorder
* Special diet preventing the low FODMAP diet
* Other GI disease or other disease explaining symptoms
* Medication intake explaining symptoms
* Not able to follow protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal symptoms | Week 8
  IBS-SSS questionnaire

SECONDARY OUTCOMES:
Change in Quality of life | Week 8
  SF-36 questionnaire
Pain diary | Daily during the study
  VAS scales on a daily basis

CONTACTS AND LOCATIONS:
Overall Officials: Anne L Krarup, PhD, Principal Investigator — Regionshospital Nordjylland; Jeanette Soerensen, PhD-student, Principal Investigator — Regionshospital Nordjylland
Locations (1):
- North Denmark Regional Hospital, Hjørring, North Denmark, Denmark